CLINICAL TRIAL: NCT07036354
Title: Evaluation of the Effects of Human-Animal Interaction on Physiological and Psychological Anxiety Markers in Graduate Students
Brief Title: Evaluation of the Effects of Human-Animal Interaction on Anxiety in Graduate Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wichita State University (Other)
Responsible Party: Principal Investigator, Nicole D Windsor, PT, DPT, PhD, FAAOMPT, Associate Teaching Professor, Wichita State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB6006
Record Dates: First submitted 2025-06-10; First posted 2025-06-25 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-06

CONDITIONS: Human-animal Interaction; Anxiety
MeSH Terms: conditions — Human-Animal Interaction; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human-Animal Interaction (Experimental)
  Interventions: Other: Human-Animal Interaction
- General Health Education (Active Comparator)
  Interventions: Other: General Health Education

INTERVENTIONS:
Other: Human-Animal Interaction — HAI - participants spend a specific amount of time with a therapy dog in a controlled environment.
  Arms: Human-Animal Interaction
Other: General Health Education — GHE - participants will be educated on strategies to assist in managing general and academic anxiety.
  Arms: General Health Education

SUMMARY:
The study's purpose is to evaluate the effects of human-animal interaction on physiological and psychological markers in graduate students.

Graduate students face significant anxiety due to demanding coursework, long hours of studying, intense academic challenges, and the pressure to excel. Chronic stress in this population can contribute to elevated anxiety levels and measurable physiological changes, such as increased heart rate and blood pressure.

Human-animal interaction (HAI) and its effect on student stress, test anxiety, and physiological markers have been studied on college campuses, largely focusing on undergraduate students. However, research investigating the impact of HAI on graduate student stress, test anxiety, and physiological markers in high-stakes programs is limited. This study will evaluate the effectiveness of repeated HAI on graduate students' physiological markers and anxiety. The results of this study will assist participants, students outside this study, and the program administrators to appreciate the immense value of a full-time therapy dog on campus, facilitating the human-animal bond in higher education.

DETAILED DESCRIPTION:
Graduate students often experience high levels of stress and anxiety due to academic demands, financial pressures, and time constraints. These stresses can stem from rigorous coursework, competitive environments, and the pressure to meet academic and personal expectations. Additionally, many students must manage part-time jobs, clinical rotations, or other academic obligations while maintaining personal relationships and responsibilities. The financial strain of student loans, tuition costs, and daily living often can add to the many plates graduate students handle. Time constraints, particularly the need to balance multiple responsibilities with limited hours in the day, frequently result in students prioritizing academics over self-care. As a result, the cumulative toll of these stressors can lead to the presentation of chronic stress and anxiety, which research has linked to increased pain sensitivity. This heightened pain sensitivity can negatively impact overall well-being and academic performance, making it more difficult for students to concentrate, remain motivated, and succeed in their programs.1

One intervention to combat these effects is human-animal interaction (HAI), which has been shown to reduce self-reported stress and anxiety scores, enhance mood, and promote relaxation.2 Additionally, HAI has also been shown to significantly reduce heart rate in participants.2 Previous research has explored the psychological benefits of HAI, but its effects on physiological measures such as pain pressure thresholds (PPT) remain unclear. PPTs are commonly used to estimate pain sensitivity, which is often heightened in individuals experiencing chronic stress and anxiety due to dysregulation of the body's stress response systems.1 Examining the relationship between anxiety and pain sensitivity through PPTs may provide insight into the potential physiological benefits of interventions such as human-animal interaction (HAI).

PPT refers to the minimum amount of pressure that induces pain in the participant and is commonly used to assess pain sensitivity.3 Pain sensitivity refers to an individual's perception of and ability to tolerate an enduring painful stimulus. Although pain is a subjective measure, it can be influenced by the individual's perception. Research has shown that if an individual's stress tolerance is low, then they are more likely to experience elevated intensity of pain.4,5 Furthermore, research shows that if an individual has experienced an adverse life experience that they are more likely to experience a heightened sensitivity and impaired regulation of stress and pain responses.6,7 This stress and anxiety can affect PPT measures, making individuals more sensitive to perceived pain, thus lowering an individual's PPT. Recent studies using cortical testing have found that pain sensitivity is also linked to activity and neurotransmitter levels in brain regions associated with pain processing.7 Elevated glutamate levels in these cortical areas, for instance, have been correlated with greater pain perception, further highlighting the connection between the brain's stress response and physical pain.7 On the other hand, relaxation techniques and positive social environments, including those with animals, may help increase PPT measurements in individuals who have stress-related anxiety.6,7 The purpose of this study is to evaluate the effects of HAI on both pain pressure thresholds and anxiety levels in graduate students. Specifically, this study aims to determine whether repeated HAI sessions influence pre- and post-intervention measures of PPT and anxiety.

Materials and Methods Participants The sample for this study will be a sample of convenience. The research project will be presented in person to graduate students at Wichita State University and followed up with an email to seek participants. Participants will be randomly placed into two groups - experimental (HAI) and control (GHE).

Informed Consent Informed consent will be read and signed by all participants prior to beginning the study. This study has been submitted to the Wichita State University Institutional Review Board for approval; status is pending as of this writing.

Animal A therapy-dog-in-training, "Ellie", will be provided by the handler for the duration of the research. Ellie is in the process of being certified through PawPartners. She has completed the proper health and behavior screenings to ensure her fitness for human-animal interaction.

Interaction Environments The HAI sessions will be held in a quiet, temperature-controlled room furnished with comfortable seating. Subjects in the experimental group will be given 60 minutes (15 minutes over 4 weeks) of unstructured interaction with Ellie. The experimental group was able to interact with Ellie in any way that they choose, including playing with a toy, playing fetch, or regular petting, if it is safe for both Ellie and the subject. The control group was given similar accommodation and focused on general health education to assist with the management of stress and anxiety. The control group was given handouts and the opportunity to engage in discussions regarding the benefits of walking, sleep hygiene, ways to recognize stress and anxiety, and different methods to deal with stress and anxiety.

Data Analysis A paired t-test will be used to analyze the data for statistically significant differences for both the HAI, within group, and GHE group, within groups. The variable analyzed by the paired t-test was self-reported anxiety scores done at the beginning and end of the study by both the experimental group and the control group. The independent variable was time, and the dependent variable was the anxiety levels measured with the GAD-7 Scale and AAS, as well as PPTs, BP, HR, and salivary cortisol.

A mixed design ANOVA was used to separately evaluate if there were statistically significant differences for both the experimental group, within group, and for the control group, within group. The measure analyzed by the repeated measures ANOVA was pain pressure threshold (PPT) testing performed once a week for 4 weeks. Data will be recorded during each testing session. The independent variable was time, split into 4 weeks, and the dependent variable was pressure values.

Two separate independent t-tests will be used to evaluate if there were statistically significant differences between the experimental and control groups in graduate students. The first measure analyzed by an independent t-test was self-reported anxiety scores for the experimental and control groups at the end of the study. The independent variable for this test was human animal interaction, and the dependent variable was self-reported anxiety scores. The second measure analyzed by an independent t-test was final pressure values at the end of the study for the experiment and the control group. The independent variable for this test was human animal interaction, and the dependent variable was pain pressure threshold values.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled and active first-year graduate students at Wichita State University,
* Between the ages of 20-35 years.

Exclusion Criteria:

* Participants diagnosed with allergies to dogs,
* Participants with a fear of dogs,
* Participants diagnosed with mental health disorders,
* Participants with on-going mental health treatment, counseling or medications,
* Participants with a known history of cardiac pathology and/or cardiac medications.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Pain pressure threshold measurement | From beginning of study to end of 4 weekly sessions of interventions
  The pain pressure threshold (PPT) is the level of pressure at which a stimulus, initially perceived as non-painful, becomes painful. It's a measure of how sensitive a tissue is to pressure and is often used in clinical settings to assess pain perception and identify potential pain-related conditions. PPT testing helps healthcare providers assess pain sensitivity, muscle tenderness, and potential underlying conditions. It's typically measured using a pressure algometer, a device that applies controlled pressure to a specific area of the body. Pressure is gradually increased on the area being tested until the subject reports that the pressure sensation changes to pain. The pressure at which the pain sensation is reported is recorded as the PPT. PPT may be measured at different locations on the body, both near and far from the area where pain is experienced. The pressure at which pain is first reported is recorded, often in units like kilopascals (kPa) or kilograms-force (kgf).
Salivatory Cortisol Levels | From beginning of study to end of 4 weekly sessions
  Salivary cortisol testing assesses free cortisol levels in saliva, which reflect the biologically active portion of cortisol in the body. Normal ranges vary based on the time of day, with higher levels in the morning and lower levels at night. Cortisol levels naturally fluctuate throughout the day, with the highest levels typically in the early morning and the lowest in the evening. Salivary cortisol levels are often measured in nanograms per milliliter (ng/mL) or nanomoles per liter (nmol/L). Saliva collection is convenient and non-invasive, making it suitable for repeated measurements and for individuals who may have difficulty with blood draws.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | Beginning of the study to end of 4 weekly sessions of interventions
  GAD-7 is primarily used for screening and assessing the severity of generalized anxiety disorder (GAD), but it also performs reasonably well in screening for other anxiety disorders like panic disorder, social anxiety disorder, and post-traumatic stress disorder. The GAD-7 can be self-administered or administered by a clinician. It's a brief questionnaire that can be easily incorporated into various settings, including primary care and research. Each of the seven questions is answered using a 4-point Likert scale (0 = not at all, 1 = several days, 2 = more than half the days, 3 = nearly every day). The scores for all seven items are summed to get a total score. Interpretation: 0-4: minimal anxiety; 5-9: mild anxiety; 10-14: moderate anxiety; 15-21: severe anxiety. The GAD-7 has demonstrated good sensitivity and specificity as a screening tool for GAD, with a sensitivity of 89% and specificity of 82% when using a cut-off score of 10 or greater.
Academic Anxiety Scale (AAS) | Beginning of study to end of 4 weekly sessions of interventions
  The Academic Anxiety Scale (AAS) is a tool used to measure the level of anxiety students experience in academic settings. Components of academic anxiety include the generalized perception of stressors, worry, emotionality, task-generated interference, and study skills deficits. The AAS is an 11-item scale that assesses how students perceive academic stressors. The scale uses a 4-point Likert-type response format, and the total score is the sum of the responses (44 maximum to 11 minimum score). Higher scores indicate higher levels of academic anxiety. The AAS can be used in research and for screening purposes to identify students who may benefit from support or interventions.
Canine Behavioral Assessment & Research Questionnaire (C-BARQ) | Beginning of the study to the end of the 4 weekly interventions
  The C-BARQ is a standardized, behavioral evaluation tool for dog owners, handlers, and professionals. The C-BARQ was originally designed to measure the prevalence and severity of behavioral problems in dogs, and that remains its primary purpose. Behavior problems are widely acknowledged to be the most important cause of premature death in companion dogs, as well as being the primary reason why dogs are surrendered to animal shelters and rescue groups. Among working dogs, behavioral problems are the single most common reason why dogs are released from training programs. The C-BARQ is a reliable and validated method for measuring behavior problems in dogs, and is calculated on a 5-point Likert scale where owners rate their dog's behavior in various situations. Higher scores generally indicate more problematic or undesirable behaviors, with some exceptions, like trainability, where higher scores are favorable. The questionnaire assesses different domains of dog behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Wichita State University, Wichita, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants will be tracked with a unique numerical identifier; all personal demographic information will be redacted. Data will be stored and shared via a repository so that others can see our data and duplicate the study if desired.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data available 02/01/2026 and available for five (5) years.
Access Criteria: Data will be available via www.figshare.com, a data repository

REFERENCES:
- [Background] Zunhammer M, Schweizer LM, Witte V, Harris RE, Bingel U, Schmidt-Wilcke T. Combined glutamate and glutamine levels in pain-processing brain regions are associated with individual pain sensitivity. Pain. 2016 Oct;157(10):2248-2256. doi: 10.1097/j.pain.0000000000000634. PMID 27649042
- [Background] Generaal E, Vogelzangs N, Macfarlane GJ, Geenen R, Smit JH, de Geus EJ, Penninx BW, Dekker J. Biological stress systems, adverse life events and the onset of chronic multisite musculoskeletal pain: a 6-year cohort study. Ann Rheum Dis. 2016 May;75(5):847-54. doi: 10.1136/annrheumdis-2014-206741. Epub 2015 Apr 22. PMID 25902791
- [Background] Abdallah CG, Geha P. Chronic Pain and Chronic Stress: Two Sides of the Same Coin? Chronic Stress (Thousand Oaks). 2017 Feb;1:2470547017704763. doi: 10.1177/2470547017704763. Epub 2017 Jun 8. PMID 28795169
- [Background] Reezigt RR, Slager GEC, Coppieters MW, Scholten-Peeters GGM. Novice assessors demonstrate good intra-rater agreement and reliability when determining pressure pain thresholds; a cross-sectional study. PeerJ. 2023 Jan 4;11:e14565. doi: 10.7717/peerj.14565. eCollection 2023. PMID 36624753
- [Background] Ein N, Li L, Vickers K. The effect of pet therapy on the physiological and subjective stress response: A meta-analysis. Stress Health. 2018 Oct;34(4):477-489. doi: 10.1002/smi.2812. Epub 2018 Jun 8. PMID 29882342
- [Background] Wyns A, Hendrix J, Lahousse A, De Bruyne E, Nijs J, Godderis L, Polli A. The Biology of Stress Intolerance in Patients with Chronic Pain-State of the Art and Future Directions. J Clin Med. 2023 Mar 14;12(6):2245. doi: 10.3390/jcm12062245. PMID 36983246

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-10-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT07036354/Prot_ICF_000.pdf